CLINICAL TRIAL: NCT05655104
Title: Effects of Couplet Care on Parents and Parent-infant Dyad in Neonatal Intensive Care Unit: Before and After Comparison Study
Brief Title: Effects of the Couplet Care in Neonatal Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Liisa Lehtonen, Professor, Turku University Hospital
Other Study IDs: CoupletCareStudy/2022
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Early Skin-to-skin Contact; Psychological Distress; Parenting; Preterm Infant
Keywords: NICU; Family centered care; Couplet care; Parent-infant closeness; Postpartum depression
MeSH Terms: conditions — Premature Birth; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Couplet Care group and their historical controls: Postintervention group: All parents enrolled in 2022-23 are classified into this group. They receive the intervention "Couplet Care."
  Pre-intervention group: All parents enrolled in 2018-19 are treated as controls. They did not receive the intervention "Couplet Care."
  Interventions: Other: Couplet Care

INTERVENTIONS:
Other: Couplet Care — In the Couplet Care model, the parents are provided access to the infant stabilisation room and encouragement for early skin-to-skin contact, mothers receive their postpartum care in the same NICU room with the infant, and fathers/partners also have a bed in the same NICU room.

SUMMARY:
This is a quasi-experimental before and after intervention study taking place in the level III NICU of Turku University Hospital in Finland to evaluate the effects of the Couplet Care, a care model which provides maternal and infant care in the same room even when intensive care of the infant is needed. The investigators will prospectively collect data after starting Couplet Care. The pre-intervention data was already collected during 2018 and 2019 as a part of the 2nd International Closeness Survey.

DETAILED DESCRIPTION:
Background: It is essential to keep newborn infants and their parents together for the well-being of both. However, the families whose infants need admission to the neonatal intensive care unit (NICU) are often separated. One of the solutions to reduce parent-infant separation is couplet care, where both mother and newborn infant receive their postpartum care in the same hospital room, even if the infant needs intensive care. However, currently only a few NICUs practice couplet care, and the scientific evidence to support implementing couplet care has been scarce. Since moving into the new hospital building in 2022, Turku University Hospital has provided "couplet care model" for all the mother-infant pairs admitted to the neonatal intensive care unit. In addition, all NICU rooms have two adult beds to accommodate both parents.

Aims: The objective of the study is to evaluate the effects of couplet care model on parent and infant well-being. The primary outcome measure is parent-infant closeness, including 1) the time from the birth to the first skin-to-skin contact (SSC) and holding, 2) the duration of parents' presence in the NICU measured for 14 days during the first three weeks, and 3) the duration of SSC and holding measured for 14 days during the first three week after the birth. The secondary outcomes are parental postpartum depressive and anxiety symptoms, parent-infant bonding, the parent-reported quality of family centered care, and breastfeeding success up to the 4 months of corrected age. In addition, factors influencing the realization of early SSC and parents' presence in the NICU are explored by interviews and questionnaires.

Methods: This is a quasi-experimental before and after intervention study taking place in a level III NICU in Turku University Hospital. The pre-intervention data was obtained from 30 families (and 40 infants) during the 2nd International Closeness Survey in 2018 and 2019. The couplet care model has been offered to all families in Turku University Hospital NICU since February 2022. The post-intervention data will be collected prospectively starting in December 2022. The families of preterm infants born before 35 weeks will be eligible for the study. The informed consent must be obtained within 6 days of life. The recruitment will continue until 30 families with a full set of data is recruited.

The duration of parental presence and the duration of SSC in the NICU will be measured using self-reported Parent-Infant Closeness Diary during a 14-day time period after recruitment in the study. Parental postpartum depressive and anxiety symptoms, mother-to-infant bonding and parent-reported quality of family centered care will be assessed by self-report questionnaires (Edinburgh Postnatal Depression Scale, State and Trait Anxiety Inventory, Japanese version of Mother-to-Infant Bonding Scale, and modified DigiFCC, respectively). In addition, parents are asked to fill in a questionnaire about breastfeeding success. The factors influencing the practice of early skin-to-skin contact and parents´ presence in the NICU will be examined by semi-structured qualitive interviews.

ELIGIBILITY:
[Family]

Inclusion Criteria:

* Families of preterm infants born below 35 weeks of gestation at Turku University Hospital

Exclusion Criteria:

* The expected duration of hospitalization is less than 3 days
* Outborn infants
* The infants are triplets or more
* The parents cannot understand the informed consent form in either Finnish, Swedish, English, or Russian
* The infant's condition is critical and survival is uncertain

[healthcare staff]

Inclusion Criteria:

* All healthcare staff who have the possibility to participate in the decision about parent-infant early skin-to-skin contact after the delivery.

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families of preterm infants born below 35 weeks of gestation at Turku University Hospital, a level III neonatal intensive care unit in Finland
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time from the birth to the first skin-to-skin contact | at 0 day of age
  The time difference (minutes) between the birth to the first skin-to-skin contact. It will be assessed for each parent. The information will be collected from parents using the questionnaire or from the medical record.
Time from the birth to the first holding | at 0 day of age
  The time difference (minutes) between the birth to the first holding. It will be assessed for each parent. The information will be collected from parents using the questionnaire or from the medical record.
Average daily duration of parents' presence in the hospital room | at 2 weeks of age
  The duration of parents' presence in the hospital room is measured for 14 days after the consent. The average time will be calculated for each parent (hours per day). The presence is recorded using the Parent-Infant Closeness Diary. This diary is a paper format and has one day per page including three items for each parent: presence, skin-to-skin contact, and holding. Mother and father respectively draw a line on the diary for these items. The start and the end times can be marked with a 5-minute accuracy. The validity of Parent-Infant Closeness Diary has already been evaluated. Parental presence is defined as being in the infant's room in the neonatal intensive care unit.
Average duration of skin-to-skin contact | at 2 weeks of age
  The duration of skin-to-skin contact is measured for 14 days after the consent. The average time per day will be calculated for each parent (minutes per day). The time of skin-to-skin contact is recorded using the Parent-Infant Closeness Diary. This diary is a paper format and has one day per page including three items for each parent: presence, skin-to-skin contact, and holding. Mother and father respectively draw a line on the diary for these items. The start and the end times can be marked with a 5-minute accuracy. The validity of Parent-Infant Closeness Diary has already been evaluated. Skin-to-skin contact is defined as the infant being held by the parent on the bare chest, with only a diaper and a cap if necessary.
Average duration of holding | at 2 weeks of age
  The duration of holding is measured for 14 days after the consent. The average time per day will be calculated for each parent (minutes per day). The time of skin-to-skin contact is recorded using the Parent-Infant Closeness Diary. This diary is a paper format and has one day per page including three items for each parent: presence, skin-to-skin contact, and holding. Mother and father respectively draw a line on the diary for these items. The start and the end times can be marked with a 5-minute accuracy. The validity of Parent-Infant Closeness Diary has already been evaluated. Holding is defined as parent holding the infant who has clothes on.

SECONDARY OUTCOMES:
Parental postpartum depressive symptoms | at 2 weeks of age, at discharge (about 2 months of age), and at 4 months of corrected age
  Parental postpartum depressive symptoms will be assessed using Edinburgh Postnatal depression scale (EPDS). It is a self-report questionnaire and comprises 10 items, each of which is scored on a four-point scale (0-3). The total score varies from a minimum of 0 to a maximum of 30, and higher scores indicating more depressive symptoms. The EPDS is analyzed as a continuous variable and also as a proportion of parents exceeding the cutoff score. The cutoff score of clinical depression is 13 or more for mothers and 10 or more for fathers.
Parental anxiety symptoms | at discharge (about 2 months of age)
  Parental anxiety symptoms will be assessed using STAI. The STAI questionnaire assesses two different anxiety types at the same time. State anxiety is an emotional response that can change over time according to the situation. Trait anxiety indicates a personal emotional characteristic that a person has. There are 20 questions for each state and trait anxiety and each is scored on a four-point scale (1-4). The total score in each type of anxiety varies from a minimum of 20 to a maximum of 80, and higher scores indicating more anxiety symptoms. The cutoff score of state anxiety usually used for a postpartum period is 40 or more: those who have a total state-STAI score of 40 or more have higher postpartum anxiety symptoms.
Parent-infant bonding | at discharge (about 2 months of age)
  The feelings of bonding felt by parent towards the newborn are assessed using the Japanese version of Mother-to-Infant Bonding Scale (MIBS-J). MIBS-J is a self-report questionnaire and comprises ten items, each of which is scored on a four-point scale (0-3). The total score varies from 0 to 30, and higher scores indicating a weaker bonding between a mother and her infant.
Quality of family centered care as reported by parents | at discharge (about 2 months of age)
  The family centered care provided by the medical professionals in the NICU is assessed by parents using a questionnaire modified from DigiFCC questions. It consists of 9 questions. Each question has the Likert scale from 1 to 7 (1 not at all and 7 very much; 0 not applicable). A higher score indicates better family centered care received by parents. The average score of all questions will be used.
  For families in the pre-intervention cohort, investigators used the same questions but they were delivered daily: parents received one out of the 9 questions as a text message in a random order every evening and responded by a score using their mobile phone.
Breastmilk feeding | at discharge (about 2 months of age) and at 4 months of corrected age
  Parents are asked a question about breastmilk feeding status: whether the infant is on only breast milk, partially on breast milk, or not on breast milk.
Breastfeeding | at discharge (about 2 months of age) and at 4 months of corrected age
  Parents are asked a question about the breastfeeding status: whether the infant is fed from the breast, bottle, feeding tube, or by any other method.

OTHER OUTCOMES:
Qualitative interviews for parents | at 2 weeks of age
  To understand the factors which influence the parental decision to stay or not to stay in the neonatal intensive care unit. The sample size will be based on data saturation, usually reached with 15-25 participants. Eligible families for the qualitative interview will be selected based on purposive sampling. Investigators aim to recruit both 1) mothers and fathers, 2) parents who stay less than 8 hours per day in the unit and parents who are in the unit almost 24/7, and 3) Finns and immigrants. Face-to-face The interviews will be conducted in Finnish or English by research nurses, neonatologists, or medical students. A suitable time will be agreed with the participants in advance. The duration of each interview will last from 30 minutes to one hour. Interviews are recorded for the purpose of the analysis. The interview guide will be pilot tested with 2-3 first participants and modified if needed.
Qualitative interviews for healthcare staff in the neonatal intensive care unit | within about a week after the decision of early skin-to-skin contact is made
  To analyze how the decision was made to conduct or not to conduct early parent-infant skin-to-skin contact. Eligible staff members for these qualitative interviews will be selected based on purposive sampling. The investigators aim to recruit the members of the multi-professional team involved in the delivery of a preterm baby. The investigators perform face-to-face interviews with the members of the team about the decision-making related to skin-to-skin contact. The interviews will be conducted in Finnish by a research nurse. The teams are informed about the interviews after the stabilization and suitable times will be planned so that one or several team members participate at a time. A semi-structured interview guide will be used. The duration of each interview will be 20-60 minutes. Interviews are recorded for the purpose of the analysis.
Questionnaire of Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) | any time during the study period, within about six months after the start of this study
  These questionnaires are used to measure the readiness for the Couplet Care intervention. Staff members will be given these three self-reported questionnaires as one questionnaire including 12 questions that are rated using a Likert scale from 1 (fully disagree) to 5 (fully agree). The measure has been shown to be valid and reliable to measure acceptability, appropriateness, and feasibility of an intervention.
Emotional Closeness questionnaire | at discharge (about 2 months of age)
  The emotional closeness scale is a self-report questionnaire to assess parents' emotional closeness to their infants who require neonatal care. The scale comprises 27 items, each of which are scored on a VAS scale (0-100 mm). The total score varies from 0 to 2700. The higher scores indicate a higher level of parental emotional closeness. The scale will be piloted in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Lehtonen, MD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No
The investigators do not have a plan to make the data open in the future. However, it can be shared with another personnel or research team for another scientific purposes with the permission of the principal investigator and any other necessary procedures.